CLINICAL TRIAL: NCT03343847
Title: A Phase 3 Randomized Placebo-controlled Double-blind Study of Romiplostim for the Treatment of Chemotherapy-induced Thrombocytopenia in Patients Receiving Chemotherapy for Treatment of Lymphomas
Brief Title: Study of Romiplostim for Chemotherapy-induced Thrombocytopenia in Adult Subjects With Lymphoma.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was not feasible
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140347; 2017-002995-16 (EudraCT Number)
Record Dates: First submitted 2017-10-12; First posted 2017-11-17 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Chemotherapy-induced Thrombocytopenia
MeSH Terms: interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Romiplostim (Experimental): the study in a 2:1 randomization ratio(108 subjects to romiplostim)
  Interventions: Biological: Romiplostim
- Placebo (Placebo Comparator): the study in a 2:1 randomization ratio (54 subjects to placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Romiplostim — This trial is designed to study romiplostim for the treatment of chemotherapy-induced thrombocytopenia (CIT) in patients receiving chemotherapy for the treatment of lymphoma.
  Arms: Romiplostim
Other: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of romiplostim for the treatment of CIT in patients receiving chemotherapy for the treatment of lymphomas measured by the ability to administer on-time, full-dose chemotherapy.

DETAILED DESCRIPTION:
This is a phase 3, randomized, placebo-controlled, multicenter, international study for the treatment of CIT in adult subjects receiving chemotherapy for the treatment of lymphomas, defined by 2 platelet counts < 30 x 10^9/L at least 7 days apart. The study will consist of a screening period of up to 4 weeks, a 16-week treatment period, an end-of-treatment (EOT) visit, and long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 101 Subject has provided informed consent/assent prior to initiation of any study-specific activities/procedures or subject's legally acceptable representative has provided informed consent prior to any study-specific activities/procedures being initiated when the subject has any kind of condition that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent.
* 102 Males or females ≥ 18 years of age at signing of the informed consent.
* 103 Documented active lymphoma.
* 104 Receiving cancer treatment with 14-, 21-, or 28-day cycles, using medication such as alkylating agents, anthracyclines, carboplatin, cisplatin, nucleoside analogs, or any other chemotherapy agents with thrombocytopenia as a warning or adverse reaction.
* 105 Subjects must have 2 platelet counts < 30 x 109/L at least 7 days apart as a result of the chemotherapy administered in the cycle immediately preceding study entry, and no platelet count ≥ 50 x 109/L during 3-week period prior to enrollment despite dose delay or dose modification of chemotherapy regimen. The first platelet count < 30 x 109/L may be collected from local lab platelet count and must be confirmed within the 28-day screening period.
* 106 Subjects must not have received chemotherapy within 14 days prior to first dose of investigational product.
* 107 Subjects must have at least 4 additional planned cycles of chemotherapy at study enrollment.
* 108 Subjects must be able to receive the same chemotherapy regimen (when possible, same schedule and same agents) for at least 2 additional cycles per investigator judgement.
* 109 Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* 201 Acute lymphoblastic leukemia.
* 202 Acute myeloid leukemia.
* 203 Any myeloid malignancy.
* 204 Myelodysplastic syndrome.
* 205 Myeloproliferative disease.
* 206 Multiple myeloma.
* 207 Within 4 months prior to enrollment, any history of active congestive heart failure (New York Heart Association [NYHA] class III to IV), symptomatic ischemia, uncontrolled arrhythmias, clinically significant electrocardiogram (ECG) abnormalities, screening ECG with corrected QT (QTc) interval of > 470 msec, pericardial disease, or myocardial infarction.
* 208 New or uncontrolled venous thromboembolism or thrombotic events within 3 months prior to screening.
* 209 Known human immunodeficiency virus infection, hepatitis C infection, or hepatitis B infection (subjects with hepatitis B surface antigen or core antibody receiving and responding to antiviral therapy directed at hepatitis B are allowed).
* 210 Secondary malignancy within the past 5 years except: Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease. Adequately treated cervical carcinoma in situ without evidence of disease. Adequately treated breast ductal carcinoma in situ without evidence of disease. Prostatic intraepithelial neoplasia without evidence of prostate cáncer. Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.

Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician (excluding malignancies listed in exclusion criteria 201 to 206).

* 211 Previous use of romiplostim, pegylated recombinant human megakaryocyte growth and development factor, eltrombopag, recombinant human TPO, any other TPO receptor agonist, or any investigational platelet producing agent.
* 212 Currently receiving treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* 213 Anemia (hemoglobin < 8 g/dL) on the day of initiation of investigational product. Use of red cell transfusions and erythropoietic stimulating agents is permitted as per institutional guidelines.
* 214 Neutropenia (absolute neutrophil count < 1 x 109/L) on the day of initiation of investigational product. Use granulocyte-colony stimulating factor is permitted as per institutional guidelines.
* 215 Abnormal renal function with serum creatinine ≥ 1.5 times [X] the upper limit of normal [ULN] OR creatinine clearance ≤ 60 mL/min using Cockcroft-Gault estimated creatinine clearance as assessed by central laboratory during screening.
* 216 Abnormal liver function (TBL > 3x ULN; alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 3x ULN for subjects without liver metastases or ≥ 5x ULN for subjects with liver metastases) as assessed by central laboratory during screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-27 (Estimated); Primary Completion 2021-07-17 (Estimated); Study Completion 2021-07-17 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy dose delay or reduction | 17 weeks
  Either a chemotherapy dose delay by
  ≥ 4 days or chemotherapy dose reduction by ≥ 15% due to thrombocytopenia as measured in any 2 planned cycles of chemotherapy during the treatment period.

SECONDARY OUTCOMES:
Platelet recovery | 7 days post transfusion through platelet recovery
  The time to first platelet recovery, defined by platelet count ≥ 50 x 10^9/L in the absence of platelet transfusions during the preceding 7 days
Platelet count | 7 days after 3rd dose of IP with no transfusions in preceding 7 days
  Achieving a platelet count
  ≥ 50 x 10^9/L, assessed 7 days after the third dose of investigational product and in the absence of platelet transfusions during the preceding 7 days
Depth of the platelet count | 3rd dose of IP through End of treatment, up to 43 months
  The depth of the platelet count nadir for chemotherapy cycles administered after the third dose of investigational product through the end of the treatment period
Subject Incidence of Platelet Transfusion | Through treatment period, up to 17 weeks
  Incidence of platelet transfusions during the treatment period
Bleeding events | Through treatment period, up to 17 weeks
  the duration-adjusted event rate of
  ≥ grade 2 bleeding events, as assessed by the Common Terminology Criteria for Adverse Events (CTCAE), during the treatment period
Adverse Events, Serious Adverse Events, clinically significant lab value changes | Through treatment period, up to 17 weeks
  adverse events, including treatment-emergent adverse events, serious adverse events and clinically significant changes in laboratory values
Antibody Formation | throughout treatment period, up to 17 weeks
  anti-romiplostim antibodies and antibodies to TPO
Vital Status | treatment period through end of study, up to 43 months
  vital status
Changes in health | treatment period through end of study, up to 43 months
  myelodysplastic syndromes and secondary malignancies

OTHER OUTCOMES:
Platelet count | treatment period through end of study, up to 43 months
  Exploratory - Percentage of time with a platelet count ≥ 50 x 10^9/L, starting after the third dose of investigational product through the end-of-treatment period, in the absence of platelet transfusions during the preceding 7 days.
Change in Clinical Outcome Assessment (COA) scores | Through treatment period, up to 17 weeks
  Change in Patient Global Assessment-CIT (PGA-CIT) scores from week 1 (baseline) to weeks 2 and 3.
  1. 4-item instrument designed to assess global change in quality of life and symptoms over time (since the previous clinic visit).
  2. The amount of change is rated using a 7-point Likert-style scale ranging from 1 (very much worse) to 7 (very much better). Items are scored as single items with higher scores indicating a greater degree of improvement.
Change in Health-Related Quality of Life (HRQoL) score | Through treatment period, up to 17 weeks
  Change in Patient Global Assessment-CIT (PGA-CIT) scores from week 1 (baseline) to weeks 2 and 3.
  1. 4-item instrument designed to assess global change in quality of life and symptoms over time (since the previous clinic visit).
  2. The amount of change is rated using a 7-point Likert-style scale ranging from 1 (very much worse) to 7 (very much better). Items are scored as single items with higher scores indicating a greater degree of improvement.
Romiplostim concentration | Through treatment period, up to 17 weeks
  Exploratory - Trough serum concentration of romiplostim
Change in Clinical Outcomes Assessment (COA) scores | Through treatment period, up to 17 weeks
  European Quality of Life-5 Dimensions (EQ-5D) scores from week 1 (baseline) to weeks 2 and 3.
  1. The EQ-5D provides a simple descriptive health profile and a single index value for health status. The EQ-5D descriptive health profile comprises 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension comprises 3 levels (no problems, some/moderate problems, extreme problems). A unique EQ-5D-3L health state is defined by combining one level from each of the 5 dimensions.
  2. EQ-5D Index values range from -0.59 to 1.00. In addition, the EQ-5D includes a single item visual analogue scale item that records the subject's self-rated health status on a vertical graduated (0 to 100) line. Higher EQ-5D index and visual analogue scale scores represent better health status.
Change in Clinical Outcomes Assessment (COA) scores | Through treatment period, up to 17 weeks
  Change in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue scores from week 1 (baseline) to weeks 2 and 3.
  Version 4 (for patients with thrombocytopenia) and 2) a patient global assessment - CIT (PGA-CIT) instrument
  1. The FACT-Th18 is a 45-item instrument that includes 28 FACT general items covering 4 domains (physical well-being, social/family well-being, emotional well-being, and functional well-being) with an additional 17 items covering Additional Concerns, 15 of which specific to thrombocytopenia.
  2. Scale scores range from 0 (Not at all) to 4 (Very Much) and can be derived for each of the 4 FACT--G domains, a FACT-G total score, a thrombocytopenia subscale score, and a FACT-Th total score. The FACT-Th has been evaluated as a reliable and valid measure for assessing the impact of thrombocytopenia on patients' lives that can distinguish cancer patients with and without thrombocytopenia and is responsive to increase in platelet count over time.
Change in Health-Related Quality of Life (HRQoL) score | Through treatment period, up to 17 weeks
  European Quality of Life-5 Dimensions (EQ-5D) scores from week 1 (baseline) to weeks 2 and 3.
  1. The EQ-5D provides a simple descriptive health profile and a single index value for health status. The EQ-5D descriptive health profile comprises 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension comprises 3 levels (no problems, some/moderate problems, extreme problems). A unique EQ-5D-3L health state is defined by combining one level from each of the 5 dimensions.
  2. EQ-5D Index values range from -0.59 to 1.00. In addition, the EQ-5D includes a single item visual analogue scale item that records the subject's self-rated health status on a vertical graduated (0 to 100) line. Higher EQ-5D index and visual analogue scale scores represent better health status.
Change in Health-Related Quality of Life (HRQoL) score | Through treatment period, up to 17 weeks
  Change in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue scores from week 1 (baseline) to weeks 2 and 3.
  Version 4 (for patients with thrombocytopenia) and 2) a patient global assessment - CIT (PGA-CIT) instrument
  1. The FACT-Th18 is a 45-item instrument that includes 28 FACT general items covering 4 domains (physical well-being, social/family well-being, emotional well-being, and functional well-being) with an additional 17 items covering Additional Concerns, 15 of which specific to thrombocytopenia.
  2. Scale scores range from 0 (Not at all) to 4 (Very Much) and can be derived for each of the 4 FACT--G domains, a FACT-G total score, a thrombocytopenia subscale score, and a FACT-Th total score. The FACT-Th has been evaluated as a reliable and valid measure for assessing the impact of thrombocytopenia on patients' lives that can distinguish cancer patients with and without thrombocytopenia and is responsive to increase in platelet count over time.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com